CLINICAL TRIAL: NCT04380545
Title: A Phase I/II Study of Nivolumab Plus 5-Fluorouracil Plus Interferon-α2b for Unresectable Fibrolamellar Hepatocellular Carcinoma
Brief Title: Nivolumab, Fluorouracil, and Interferon Alpha 2B for the Treatment of Unresectable Fibrolamellar Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1135; NCI-2020-02614 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1135 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stage III Hepatocellular Carcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Unresectable Fibrolamellar Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorouracil; dehydroftorafur; Nivolumab; recombinant interferon alpha 2b-like protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (fluorouracil, interferon alpha 2b, nivolumab) (Experimental): Patients receive fluorouracil IV continuously on days 1-7 and 15-21 and recombinant interferon alpha 2b-like protein SC on days 1, 3, 5, 15, 17, and 19. Treatment repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 3, patients receive nivolumab IV over 30 minutes on day 1, fluorouracil IV continuously on days 1-7 and 15-21, and recombinant interferon alpha 2b-like protein interferon alpha 2b SC on days 1, 3, 5, 15, 17, and 19. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Biological: Nivolumab; Biological: Recombinant Interferon Alpha 2b-like Protein

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: Recombinant Interferon Alpha 2b-like Protein — Given SC
  Other Names: Novaferon; Recombinant IFN Alfa-2b-like Protein

SUMMARY:
This phase I/II trial studies the side effects and how well nivolumab, fluorouracil, and interferon alpha 2b work for the treatment of fibrolamellar cancer (liver cell cancer) that cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Interferon alpha 2b may help stimulate the immune system to fight cancer. Giving nivolumab, fluorouracil, and interferon alpha 2b may work better in treating unresectable fibrolamellar cancer compared to fluorouracil and interferon alpha 2b alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of therapy with nivolumab + fluorouracil (5-FU) + recombinant interferon alpha 2b-like protein (IFN-alpha2b) in patients with unresectable fibrolamellar hepatocellular carcinoma (FLHCC) in the context of palliative systemic and prebiopsy therapy.

SECONDARY OBJECTIVE:

I. To assess the efficacy of nivolumab + 5-FU + IFN-alpha2b therapy in patients with unresectable FLHCC by estimating the overall response rate (ORR) and progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, and comparing those rates to those from historical controls in our published data.

EXPLORATORY OBJECTIVES:

I. To assess the immunological/biomarker changes in tumor tissues and peripheral blood in response to nivolumab + 5-FU + IFN-aplha2b therapy (pre- versus [vs] post-treatment).

II. To explore any potential association between these biomarker measures and both antitumor response and immune-related response criteria (irRC) assessed by the University of Texas MD Anderson Cancer Center (MD Anderson) Department of Diagnostic Imaging.

OUTLINE:

Patients receive fluorouracil intravenously (IV) continuously on days 1-7 and 15-21 and recombinant interferon alpha 2b-like protein subcutaneously (SC) on days 1, 3, 5, 15, 17, and 19. Treatment repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning in cycle 3, patients receive nivolumab IV over 30 minutes on day 1, fluorouracil IV continuously on days 1-7 and 15-21, and recombinant interferon alpha 2b-like protein interferon alpha 2b SC on days 1, 3, 5, 15, 17, and 19. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients, or their legal guardian, must give written informed consent prior to initiation of therapy, and patients under age 18 must give assent in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy
* Patients with histologically confirmed FLHCC (or with documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable). The determination of resectability status will ultimately lie in the clinical judgment of the surgical oncologist and medical oncologist involved in the care of the patient. The definition of resectability is as follows: hepatectomy can achieve a negative margin while preserving more than 30% of the total estimated liver volume, sparing two contiguous hepatic segments, and maintaining vascular inflow, vascular outflow, and biliary drainage. Patients with extrahepatic disease are defined as having unresectable disease
* Patient must have measurable disease defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures >= 15 mm with conventional techniques or >= 10 mm with more sensitive techniques such as magnetic resonance imaging (MRI) or spiral computed tomography (CT) scan
* Eastern Cooperative Oncology Group performance status (ECOG PS =< 1), or for patients under age 18 Karnofsky performance status of >= 70
* No advanced cirrhosis, with Child-Pugh A
* Absolute neutrophil count (ANC) >= 1,000 /mm^3 (within 14 days of the first dose of study drug)
* Platelets >= 100,000 /mm^3 (within 14 days of the first dose of study drug)
* Hemoglobin > 9.0 g/dL (may be transfused or receive epoetin alfa [e.g., Epogen] to maintain or exceed this level) (within 14 days of the first dose of study drug)
* Total bilirubin =< 1.5 mg/dL (within 14 days of the first dose of study drug)
* Serum creatinine =< 1.5 times the upper limit of normal (ULN) or estimated creatinine clearance (CrCL) > 40 mL/min (within 14 days of the first dose of study drug)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 times institutional ULN (within 14 days of the first dose of study drug)
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study drug
* Women must not be breastfeeding
* WOCBP must agree to follow instructions for method(s) of contraception from the time of enrollment for the duration of treatment with study drug(s) plus 5 half-lives of study drug(s) plus 30 days (duration of ovulatory cycle) for a total of 5 months post treatment completion
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug(s) plus 90 days (duration of sperm turnover) for a total of 7 months post-treatment completion
* Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing as described in these sections. Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception, which have a failure rate of < 1% per year when used consistently and correctly. At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below:

  * HIGHLY EFFECTIVE METHODS OF CONTRACEPTION:

    * Male condoms with spermicide
    * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices such as Mirena by WOCBP subject or male subject's WOCBP partner
    * Nonhormonal intrauterine devices, such as ParaGard
    * Tubal ligation
    * Vasectomy
    * Complete Abstinence

      * Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Abstinence is only acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, profession of abstinence for entry into a clinical trial, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence
  * LESS EFFECTIVE METHODS OF CONTRACEPTION:

    * Diaphragm with spermicide
    * Cervical cap with spermicide
    * Vaginal sponge
    * Male condom without spermicide
    * Progestin-only pills by WOCBP subject or male subject's WOCBP partner
    * Female condom

      * A male and female condom must not be used together

Exclusion Criteria:

* Any other malignancy from which the patient has been disease-free for less than 2 years, except for non-melanoma skin cancer, or in situ carcinoma of any site
* Patients who have organ allografts
* Patients who have had a major surgical procedure, open biopsy, or significant traumatic injury with poorly healed wound within 6 weeks prior to first dose of study drug; or have an anticipated need for major surgical procedure during the course of the study (other than defined by protocol). NOTE: Patients will be allowed to start cycle 1 day 1 therapy after 24 hours from pre-treatment biopsy
* Autoimmune disease: patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis])
* Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome
* Any underlying medical condition, which in the opinion of the investigator will make the administration of study drug hazardous or will obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* Patients who have had a history of acute diverticulitis, abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, gastrointestinal obstruction, or abdominal carcinomatosis which are known risks factors for bowel perforation
* Patients who have a primary brain tumor (excluding meningiomas and other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of stroke within the past year
* History of serious systemic disease, including myocardial infarction or unstable angina within the last 12 months, history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (blood pressure of > 140/90 mmHg) at the time of enrollment, New York Heart Association grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), or significant vascular disease or symptomatic peripheral vascular disease
* Patients who have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Patients who have received any live or attenuated viral vaccines within a month prior to initiation of study drugs
* Patients who have active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening

  * Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test and negative HBV deoxyribonucleic acid (DNA) test at screening, are eligible for the study
* Patients who have active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV ribonucleic acid (RNA) test at screening

  * The HCV RNA test will be performed only for patients who have a positive HCV antibody test
* Patients who have clinical history of coagulopathy, bleeding diathesis, or thrombosis within the past year
* Patients who have a serious, non-healing wound, ulcer, or bone fracture
* Patients who are pregnant (positive pregnancy test) or lactating
* Patients with prior orthotropic liver transplantation
* Patients with cirrhosis and severe synthetic liver dysfunction (Child Pugh B-C)
* Patients must not have received prior anticancer therapy with anti-PD-1 for FLHCC treatment. Patients receiving any concomitant systemic therapy for FLHCC are excluded
* Patients must not be scheduled to receive another experimental drug while on this study
* Patients who require ongoing anticoagulation will be excluded. Only aspirin will be permitted. Pre and post-surgical prophylactic anti-coagulation treatment is permitted
* Patients must not require total parenteral nutrition
* Patients who are on high dose steroid (e.g. > 10 mg prednisone daily or equivalent) or other more potent immune suppression medications (e.g. infliximab). Corticosteroid use will only be allowed during trial participation for grade 3/4 AEs or hypersensitivity reactions
* Any patients who cannot be compliant with the appointments required in this protocol must not be enrolled in this study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last treatment dose
  Safety will be monitored by addressing and recording all adverse events (AEs), serious adverse events (SAEs) and specific laboratory abnormalities (worst grade). Toxicities will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 weeks after initiation of combined treatment
  Overall response rate (ORR) is defined as the number of subjects with the best response of complete response (CR) or partial response (PR) (by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) divided by the number of subjects who started treatment.
Conversion rate to surgery | Up to 6 years
  Conversion rate to surgery is defined as the proportion of patients that will be able to receive surgery after the initiation of the study treatment divided by the number of subjects who started treatment. The conversion rate to surgery will be estimated along with the 95% confidence interval (CI).
Progression-free survival (PFS) | From the start of treatment to date of patient death (PD), to date of last follow-up if patient is alive without PD, or to date of death, whichever occurs first, assessed up to 6 years
  The Kaplan-Meier method will be used to estimate probability of PFS.

OTHER OUTCOMES:
Tissue and blood immunohistochemistry | Pre-treatment, 8 weeks, and time of discontinuation
  Each tumor will be immuno-profiled using flow cytometry (CyTOF) and immunohistochemistry (IHC). Immune responses, such as infiltration of CD8+/CD4+ T cells and dendritic cells, and cytokine levels in blood, will be compared between pre-treatment and post-treatment via paired t-test and Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Sunyoung Lee, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] O'Neill AF, Church AJ, Perez-Atayde AR, Shaikh R, Marcus KJ, Vakili K. Fibrolamellar carcinoma: An entity all its own. Curr Probl Cancer. 2021 Aug;45(4):100770. doi: 10.1016/j.currproblcancer.2021.100770. Epub 2021 Jul 1. PMID 34272087
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org